CLINICAL TRIAL: NCT02629198
Title: The Effect of Body Weight on Vitamin D Metabolism
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Department of Health, United Kingdom (Other Government); University of Sheffield (Other); MRC Human Nutrition Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: STH16353
Record Dates: First submitted 2015-12-07; First posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Osteoporosis; Obesity
Keywords: Vitamin D
MeSH Terms: conditions — Osteoporosis; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, plasma, urine, DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- normal weight: Healthy men and women ages 25-40 and 55-75. BMI 18.5 to 25.0
- overweight: Healthy men and women ages 25-40 and 55-75. BMI 25.0 to 30.0
- obese: Healthy men and women ages 25-40 and 55-75. BMI over 30

SUMMARY:
There is current interest in the role of vitamin D in the prevention and treatment of many chronic diseases, including osteoporosis, cancer and neurological disease. The majority of vitamin D in the UK comes from the action of sunlight on skin, and very little from dietary sources. Half of the adult United Kingdom (UK) population have vitamin D insufficiency (according to the Institute of Medicine definition). There are still several important unknowns, including what the optimum levels of vitamin D are, and whether the same intake of vitamin D is appropriate for all sections of the population.

Low 25(OH)D and high parathyroid hormone (PTH) have been observed in people with high adiposity (obesity), and the summer rise in vitamin D is blunted in obesity. The potential causes of low 25(OH)D levels include an inadequate supply of vitamin D (by reduced sunlight exposure or poor nutrition), the large pool size of adipose tissue or increased metabolic clearance rate.

The investigators will measure metabolites of vitamin D and the kinetics of 25(OH)D using stable isotope techniques in lean, overweight and obese men, women and children to establish whether age, gender and obesity affect vitamin D metabolism and clearance rate.

If low 25(OH)D in obesity is related to poorer skeletal health and is due to increased clearance of 25(OH)D or large pool size, then total requirements, and hence supplementation requirements, would be larger for obese people than for lean people.

DETAILED DESCRIPTION:
Part 1: Measurement of vitamin D and metabolites (adults and children) Circulating levels of vitamin D metabolites are influenced by calcium intake, so participants will be asked to complete a seven day diet diary before the first vitamin D measurement. Measured vitamin D is influenced by vitamin D binding protein, lipids and inflammatory cytokines, so the investigators will include and correct for these measurements.

Visit 1 Consent Height and weight Diet diary instructions Urine collection instructions

Visit 2 Return of 24h urine collection for calcium and creatinine Return of diet diary Fasting blood sample for vitamin D, binding protein and metabolites C reactive protein (CRP), lipids and creatine kinase (CK), PTH, insulin-like growth factor -1 (IGF-1), creatinine, calcium, albumin, phosphate

Part 2: Measurement of vitamin D clearance rate (adults only) Kinetic studies will be perturbed by acute changes in vitamin D (most likely to be caused by sunlight exposure on a sunny day), and so the studies will all be conducted in the autumn, winter, and early spring when sunlight in Sheffield will not be strong enough to deliver large doses of vitamin D.

The administration and sampling protocol for the kinetics study has been developed by statisticians at the Sheffield School of Health and Related Research (ScHaRR) in collaboration with the Medical Research Council Human Nutrition Unit, based on modelling from their previous use of the stable isotope tracer method.

Visit 2 Oral administration of stable vitamin D isotope

Visit 3 (5-7 days after visit 2) Blood sample for tracer and vitamin D metabolites

Visit 4 (9 days ± 2 after visit 2) Blood sample for tracer and vitamin D metabolites

Visit 5 (27 days ± 2 after visit 2) Blood sample for tracer and vitamin D metabolites

Visit 6 (30 days ± 2 after visit 2) Blood sample for tracer and vitamin D metabolites Height and weight

The effect of obesity on vitamin D metabolites will be determined by regression models of BMI and vitamin D measurements corrected for age and gender.

The effects of obesity on vitamin D kinetics will be determined by modelling metabolic clearance rate on age, gender and BMI.

Subjects' previous data from the 'Effects of obesity on bone structure and strength'study (STH 15688) and the 'Body weight and bone' study (STH16199) will be used to evaluate relationships between vitamin D metabolism and body fat distribution, bone density and structure, and bone biochemistry.

ELIGIBILITY:
Inclusion Criteria:

Caucasian

BMI of 18.5 kg/m2 or above for adults, 2nd-91st centile or above 98th centile for children

Ages 8 to 15 (children), 16 to 42 years (and premenopausal if female) or 55 to 77 years (and postmenopausal (at least 5 years since last menstrual period (LMP) if female)

Able and willing to participate in the study and provide written informed consent Completed either STH15688 or STH16199 and gave consent to be approached about future studies

Exclusion Criteria:

History of any long term immobilization (duration greater than three months)

Current confirmed or possible pregnancy (urinary pregnancy test if LMP >28 days)

Previously-diagnosed diabetes mellitus

History of or current conditions known to affect bone metabolism, including

* Diagnosed skeletal disease
* Chronic renal disease
* Malabsorption syndromes
* Diagnosed endocrine disorders
* Hypocalcemia or hypercalcemia
* Diagnosed restrictive eating disorder Use of medications or treatment known to affect bone metabolism, including
* Depot medroxyprogesterone or the combined oral contraceptive pill

Alcohol intake of greater than 21 units per week

Competitive athlete, defined as participating in competitive sport at amateur or professional level

Holiday with significant sunlight exposure in the last six weeks

Ages: 8 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The total study sample will consist of 136 participants (112 adults and 24 children) who are lean, overweight or obese. Participants will be drawn from two previous studies; 'The effects of obesity on bone structure and strength' (STH 15688) and 'Body weight and bone' (STH16199), in which their body composition, bone strength and biochemistry have been documented in detail.
  All participants from the previous studies will be invited to participate, and recruitment will continue until 112 adults and 24 children across a range of body weights have been recruited.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
difference in serum 25OHD between groups | one measurement at study entry (cross-sectional study)

SECONDARY OUTCOMES:
difference in 25OHD half-life between groups using the stable isotope tracer method | one measurement at study entry (cross-sectional study)
  stable isotope tracer method
difference in mean sunlight exposure score between groups (questionnaire) | one measurement at study entry (cross-sectional study)
  annual and summer sunlight score from questionnaire
difference in mean dietary vitamin D intake between groups (diet diary) | one measurement at study entry (cross-sectional study)
  habitual daily vitamin D dietary intake from diet diary
difference in mean of other serum vitamin D metabolites and measures between groups | one measurement at study entry (cross-sectional study)
  free 25OHD, 1,25OHD, vitamin D binding protein (DBP)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Walsh, MBChB PhD, Principal Investigator — University of Sheffield

IPD SHARING:
Plan to Share IPD: No